CLINICAL TRIAL: NCT01618968
Title: Exposure, Safety and Local Tolerance Study Comparing the Relative Bioavailability of Oral Methotrexate and the VIBEX™ MTX Device in Adult Subjects With Rheumatoid Arthritis
Brief Title: Comparison of Methotrexate (MTX) and the VIBEX™ MTX Device
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MTX-11-003
Record Dates: First submitted 2012-06-04; First posted 2012-06-14 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg Methotrexate (MTX) (Experimental): MTX dose group was assigned based on the subject's current therapeutic regimen of MTX and rheumatoid arthritis disease status. The sequence of treatments A, B and C was randomly assigned.
  Interventions: Drug: MTX
- 15 mg MTX (Experimental): MTX dose group was assigned based on the subject's current therapeutic regimen of MTX and rheumatoid arthritis disease status. The sequence of treatments A, B and C was randomly assigned.
  Interventions: Drug: MTX
- 20 mg MTX (Experimental): MTX dose group was assigned based on the subject's current therapeutic regimen of MTX and rheumatoid arthritis disease status. The sequence of treatments A, B and C was randomly assigned.
  Interventions: Drug: MTX
- 25 mg MTX (Experimental): MTX dose group was assigned based on the subject's current therapeutic regimen of MTX and rheumatoid arthritis disease status. The sequence of treatments A, B and C was randomly assigned.
  Interventions: Drug: MTX

INTERVENTIONS:
Drug: MTX — * Treatment A - 1 dose (4, 6, 8 or 10 tablets respectively to make up 10 mg, 15 mg, 20 mg or 25 mg MTX - per subject's dose group)
  * Treatment B - SC injection using VIBEX MTX device into abdomen (VIBEX MTX device pre-filled with 10 mg, 15 mg, 20 mg or 25 mg MTX)
  * Treatment C - SC injection using VIBEX MTX device into thigh (VIBEX MTX device pre-filled with 10 mg, 15 mg, 20 mg or 25 mg MTX)
  Other Names: Commercially available 2.5 mg MTX oral tablets; VIBEX MTX

SUMMARY:
Relative Bioavailability Comparison study

DETAILED DESCRIPTION:
A Phase 2, Open-Label, Randomized, 3-Way Crossover Study to Compare the Relative Bioavailability of Oral Methotrexate and the VIBEX™ MTX Device in Adult Subjects With Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age, diagnosed with Rheumatoid Arthritis

Exclusion Criteria:

* Pregnant females
* Any other clinically significant disease or disorder which, in the opinion of the investigator might put the subject at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Kivitz, MD;CPI, Principal Investigator — Altoona Center for Clinical Research
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

REFERENCES:
- [Derived] Schiff MH, Jaffe JS, Freundlich B. Head-to-head, randomised, crossover study of oral versus subcutaneous methotrexate in patients with rheumatoid arthritis: drug-exposure limitations of oral methotrexate at doses >/=15 mg may be overcome with subcutaneous administration. Ann Rheum Dis. 2014 Aug;73(8):1549-51. doi: 10.1136/annrheumdis-2014-205228. Epub 2014 Apr 12. PMID 24728329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 4 sites in the US. Approximately equal number of subjects on 10 mg, 15 mg, 20 mg and 25 mg doses were recruited. The dose group was determined by the Investigator based on subject's current therapeutic regimen of MTX and disease status. The subject's dose was the same for the entire study
Pre-assignment Details: MTX was administered via randomized sequence and crossover of Treatment A, Treatment B and Treatment C within the same dose group. Treatments were administered at a 7 day interval (On study days 1, 8 and 15)
Groups:
- 10mg MTX; 15mg MTX; 20mg MTX; 25mg MTX: [administered via randomized sequence and crossover of Treatment A - Oral Methotrexate (MTX) Tablets, Treatment B - SC injection of Vibex MTX into the Abdomen and Treatment C - SC injection of Vibex MTX into the Thigh]
Period: Overall Study
Arm/Group | 10mg MTX | 15mg MTX | 20mg MTX | 25mg MTX
Started | 13 | 12 | 12 | 12
Received Treatment A | 12 | 12 | 12 | 11
Received Treatment B | 13 | 12 | 12 | 12
Received Treatment C | 12 | 12 | 12 | 11
Completed | 12 | 12 | 12 | 11
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: In total, 50 subjects were randomized, of which 49 were included in the safety population. Of 49, 47 completed the study and 2 discontinued from the study after first dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | 10mg MTX | 15mg MTX | 20mg MTX | 25mg MTX | Total
Number analyzed (Participants) | 13 | 12 | 12 | 12 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.51) | 63.4 (7.49) | 60.0 (10.40) | 59.0 (11.53) | 61.4 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 8 | 7 | 31
  Male | 2 | 7 | 4 | 5 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 11 | 10 | 11 | 44
  African American | 1 | 1 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 12 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Dose-Normalized AUC[0-Inf] for MTX
Description: Dose-normalized area under the curve from time zero to infinity (AUC[0-inf]/Dose) for each treatment
Time Frame: 24 Hour period
Population: The Population was defined as all randomized subjects who received at least 1 dose of study drug and who had at least 1 valid post-dose plasma concentration value.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Groups:
- Treatment A: Oral Methotrexate (MTX) Tablets
- Treatment B: SC injection of Vibex MTX into the Abdomen
- Treatment C: SC injection of Vibex MTX into the Thigh
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 47 | 49 | 47
ng*hr/mL/mg | 109.47 (39.19) | 140.84 (46.66) | 136.45 (46.675)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; To compare the relative bioavailability of methotrexate (MTX) following oral administration to that obtained after subcutaneous (SC) injection into the abdomen using the VIBEX MTX device by measuring the area under the curve from time zero to the last measurable concentration AUC(0-inf); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference Ratio = 127.99, 90% CI 2-sided [121.61 to 134.70]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; To compare the relative bioavailability of MTX following oral administration to that obtained after SC injection into the thigh using the VIBEX MTX device by measuring the AUC(0-Inf); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference Ratio = 125.48, 90% CI 2-sided [119.43 to 131.84]
Statistical Analysis 3: Comparison: Treatment B vs Treatment C; To compare the relative bioavailability of MTX following SC injection into the abdomen to that obtained after SC injection into the thigh using the VIBEX MTX device by measuring the AUC(0-inf); Test type: Non-Inferiority or Equivalence — Test of bioequivalence was performed at each dose level; Test / Reference ratio = 101.85, 90% CI 2-sided [99.41 to 104.36]

2. Primary Outcome: Dose-Normalized AUC[0-24] for MTX
Description: Dose-normalized area under the curve from time zero to 24 hours (AUC[0-24]/Dose) for each treatment
Time Frame: 24 Hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 47 | 49 | 47
ng*hr/mL/mg | 107.64 (37.732) | 137.88 (44.513) | 133.78 (44.406)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; To compare the relative bioavailability of methotrexate (MTX) following oral administration to that obtained after subcutaneous (SC) injection into the abdomen using the VIBEX MTX device by measuring the area under the curve from time zero to the 24 hour concentration AUC(0-24); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference Ratio = 127.65, 90% CI 2-sided [121.28 to 134.36]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; To compare the relative bioavailability of methotrexate (MTX) following oral administration to that obtained after subcutaneous (SC) injection into the thigh using the VIBEX MTX device by measuring the area under the curve from time zero to the 24 hour concentration AUC(0-24); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference ratio = 125.20, 90% CI 2-sided [119.16 to 131.55]
Statistical Analysis 3: Comparison: Treatment B vs Treatment C; To compare the relative bioavailability of MTX following SC injection into the abdomen to that obtained after SC injection into the thigh using the VIBEX MTX device by measuring the area under the curve from time zero to the 24 hour concentration AUC(0-24); Test type: Non-Inferiority or Equivalence — Test of bioequivalence was performed at each dose level; Test / Reference Ratio = 101.82, 90% CI 2-sided [99.39 to 104.31]

3. Primary Outcome: Dose-Normalized Cmax for MTX
Description: Dose-normalized maximum observed concentration (Cmax) for each treatment
Time Frame: 24 Hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 47 | 49 | 47
ng/mL/mg | 22.697 (7.496) | 21.935 (8.243) | 18.436 (5.321)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; To compare the relative bioavailability of methotrexate (MTX) following oral administration to that obtained after subcutaneous (SC) injection into the abdomen using the VIBEX MTX device by measuring the maximum observed concentration (Cmax); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference ratio = 94.83, 90% CI 2-sided [86.42 to 104.06]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; To compare the relative bioavailability of methotrexate (MTX) following oral administration to that obtained after subcutaneous (SC) injection into the thigh using the VIBEX MTX device by measuring the maximum observed concentration (Cmax); Test type: Non-Inferiority or Equivalence — Bioavailability comparisons were performed at each dose level; Test / Reference Ratio = 82.12, 90% CI 2-sided [76.16 to 88.55]
Statistical Analysis 3: Comparison: Treatment B vs Treatment C; To compare the relative bioavailability of MTX following SC injection into the abdomen to that obtained after SC injection into the thigh using the VIBEX MTX device by measuring the maximum observed concentration (Cmax); Test type: Non-Inferiority or Equivalence — Test of bioequivalence was performed at each dose level; Test / Reference Ratio = 115.63, 90% CI 2-sided [108.83 to 122.86]

ADVERSE EVENTS:
Time Frame: The Safety Population was defined as all randomized subjects who received at least 1 dose of study drug. The Safety Population included 49 subjects.
Description: Adverse events were classified by treatment at onset. Any adverse event that occurred on Day 1 (after check-in) for a given treatment period was assigned to the treatment for that period.
Arm/Group | 10mg MTX | 15mg MTX | 20mg MTX | 25mg MTX
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 2/13 | 0/12 | 1/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10mg MTX (N=13) | 15mg MTX (N=12) | 20mg MTX (N=12) | 25mg MTX (N=12)
Sick Sinus Syndrome (15 mg Vibex MTX SC Thigh) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (25 mg Vibex MTX SC Abdomen) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10mg MTX (N=13) | 15mg MTX (N=12) | 20mg MTX (N=12) | 25mg MTX (N=12)
Nausea (20 mg MTX Oral) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (10 mg Vibex MTX SC Thigh) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid Arthritis (10 mg Vibex MTX SC Abdomen) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less